CLINICAL TRIAL: NCT02967731
Title: An Exploratory Safety Study of 480 Biomedical Sinus Drug Depot in Adult Subjects With Chronic Sinusitis
Brief Title: 480 Biomedical Sinus Drug Depot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lyra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 480MFSDD2016-001
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2017-06

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 480 Mometasone Furoate Sinus Drug Depot (Experimental): 480 Mometasone Furoate Sinus Drug Depot
  Interventions: Drug: 480 Mometasone Furoate Sinus Drug Depot

INTERVENTIONS:
Drug: 480 Mometasone Furoate Sinus Drug Depot — Management of Chronic Sinusitis

SUMMARY:
This is a Phase I, exploratory safety study of the 480 Biomedical Mometasone Furoate Sinus Drug Depot in adult subjects with chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CS.
* Female study subjects of child-bearing potential must have a negative pregnancy test and must agree to not become pregnant during the course of the study.
* The study subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the ethics committee of the respective clinical site.
* The study subject agrees to comply with all study requirements

Exclusion Criteria:

* Known history of intolerance to corticosteroids.
* Oral-steroid dependent condition.
* Having had corticosteroids with potential systemic effect (e.g., oral, parenteral, or high dose topical) 1 month prior to screening visit.
* Subjects with acute or chronic intracranial or orbital complications of chronic rhinosinusitis (e.g., brain abscess, related problems with eyes or central nervous system).
* Known history of hypothalamic pituitary adrenal (HPA) axial dysfunction or having morning serum cortisol level at screening outside of normal range.
* Previous pituitary or adrenal surgery.
* History or diagnosis (in either eye) of glaucoma, ocular hypertension, or cataracts.
* Recent participation in another clinical trial within 1 month of screening visit.
* Subjects currently participating in an investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Product related serious adverse events from baseline visit to 4 weeks post procedure | 4 weeks post procedure

SECONDARY OUTCOMES:
Plasma Mometasone Furoate concentration level from pre-treatment to end of treatment | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - The Queen Elizabeth Hospital, Adelaide
  - Royal Brisbane and Women's Hospital, Brisbane
  - Monash Medical Center, Melbourne
- University of Auckland, Auckland, New Zealand

REFERENCES:
- [Derived] Douglas RG, Psaltis AJ, Rimmer J, Kuruvilla T, Cervin A, Kuang Y. Phase 1 clinical study to assess the safety of a novel drug delivery system providing long-term topical steroid therapy for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Apr;9(4):378-387. doi: 10.1002/alr.22288. Epub 2019 Jan 15. PMID 30645028